CLINICAL TRIAL: NCT04291521
Title: Prospective Study of Induction Medications Used in the Rapid Sequence Intubation of Trauma Patients and a Comparison of Effects on Outcomes
Brief Title: Prospective Study of Induction Medications Used in the Trauma RSI
Acronym: ProTIM
Status: Not yet recruiting | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: University of California, Irvine (Other); University of Texas (Other); University of Chicago (Other); Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Catherine Kuza, MD, Assistant Professor, University of Southern California
Other Study IDs: HS-20-00328
Record Dates: First submitted 2020-02-26; First posted 2020-03-02 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Trauma; Rapid Sequence Intubation
Keywords: trauma; induction medications; rapid sequence intubations; outcomes
MeSH Terms: conditions — Wounds and Injuries | interventions — Ketamine; Etomidate; Propofol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult trauma patients requiring RSI: Patients who received an induction medication for intubation.
  Interventions: Drug: Ketamine; Drug: Etomidate; Drug: Propofol

INTERVENTIONS:
Drug: Ketamine — Administering ketamine as an induction medication for intubating adult trauma patients within 24 hours of hospital admission.
  Other Names: Ketalar
Drug: Etomidate — Administering etomidate as an induction medication for intubating adult trauma patients within 24 hours of hospital admission.
  Other Names: Amidate
Drug: Propofol — Administering propofol as an induction medication for intubating adult trauma patients within 24 hours of hospital admission.
  Other Names: Diprivan

SUMMARY:
To compare the outcomes of the use of propofol, etomidate, and ketamine as induction agents for adult trauma patients undergoing intubation within 24 hours of admission. The primary goal is to determine the ideal agent that should be used in this patient population for intubations.

DETAILED DESCRIPTION:
Rationale:

Although rapid sequence intubation (RSI) is commonly used in the emergency department (ED) or operating room (OR) for trauma patients, there is not one induction medication which has been deemed the drug of choice for this particular use. There is a wide variation in induction agents used by providers performing RSIs, including propofol, ketamine, methohexital, midazolam, fentanyl, and etomidate. However, no society guidelines exist on the induction agent of choice in trauma for either hemodynamically stable or unstable patients. The purpose of this study is to compare the effects of 3 of the most commonly used induction agents (propofol, etomidate, and ketamine) for RSIs in adult trauma patients on outcomes, such as mortality, and hemodynamic status. Ultimately, the investigators would like to lay the groundwork for developing guidelines that define the ideal induction agent for trauma RSIs.

Intervention: Giving propofol, ketamine, or etomidate as the induction medication for a rapid sequence intubation in trauma patients requiring intubation within 24 hours of admission.

Objectives/Purpose: The purpose of this study is to compare the effects of 3 of the most commonly used induction agents (propofol, etomidate, and ketamine) for RSIs in adult trauma patients on outcomes such as mortality. Additionally, how each agent effects patients' hemodynamic status will be evaluated. Additional outcomes of these medications will be studied in three subsets of patients: 1. those with traumatic brain injuries, 2. elderly patients (>=65-years-old), and 3. those with a low shock index (<0.9) compared to a high shock index (>0.9). Finally, the practices and outcomes of RSIs performed in the ED versus the OR will be compared. Ultimately, the investigators would like to lay the groundwork for developing guidelines that define the ideal induction agent for trauma RSIs.

Study population: Adult trauma patients undergoing RSI within 24 hours of hospital admission

Methodology: A multicenter, prospective observational study will be performed.

Endpoints: In-hospital mortality, 28-day mortality, ICU and total hospital length of stay, complications, hypotension and vasopressor use 30 minutes and 24 hours after intubation, mechanical ventilator days, and discharge disposition

Statistic plan: Data will be entered into a password-protected online data collection tool known as RedCap, and analyzed using SAS version 9.4 (SAS Institute, Inc., Cary, NC).

ELIGIBILITY:
Inclusion Criteria:

* Trauma patients >=18 yo requiring intubation within 24 hours of admission in either the ED or OR
* Patients received propofol, etomidate, or ketamine for induction agent

Exclusion Criteria:

* Patients who were intubated without induction agent medications
* Patients intubated outside of the hospital or in the field
* Patients who were intubated with an induction agent other than etomidate, ketamine, or propofol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult trauma patients requiring intubation within 24 hours of hospital admission.
Sampling Method: Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
in-hospital mortality | through study completion, an average of 1 year
  mortality

SECONDARY OUTCOMES:
total hospital length of stay | through study completion, an average of 1 year
  days
intensive care unit length of stay | through study completion, an average of 1 year
  days
mechanical ventilator days | through study completion, an average of 1 year
  days
Number of participants with hypotension | 30 minutes after intubation
  defined as systolic blood pressure<90 mmHg or mean arterial pressure <50 mmHg
Number of participants with hypotension | 24 hours after intubation
  defined as systolic blood pressure<90 mmHg or mean arterial pressure <50 mmHg
Number of participants requiring vasopressor use | 30 minutes after intubation
  vasopressor use
Number of participants requiring vasopressor use | 24 hours post intubation
  vasopressor use
number of complications | through study completion, an average of 1 year
  examples: adrenal insufficiency, aspiration, pneumonia, acute respiratory distress syndrome, organ failure, etc.
28-day mortality | 28 days after admission
  28 day mortality
discharge disposition | through study completion, an average of 1 year
  examples: discharge home no services, home with services, skilled nursing facility, rehabilitation center, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine M Kuza, MD, Principal Investigator — Keck School of Medicine of the University of Southern California
Locations (1):
- Keck School of Medicine of the University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Banh KV, James S, Hendey GW, Snowden B, Kaups K. Single-dose etomidate for intubation in the trauma patient. J Emerg Med. 2012 Nov;43(5):e277-82. doi: 10.1016/j.jemermed.2012.02.027. Epub 2012 May 3. PMID 22560133
- [Background] Jabre P, Combes X, Lapostolle F, Dhaouadi M, Ricard-Hibon A, Vivien B, Bertrand L, Beltramini A, Gamand P, Albizzati S, Perdrizet D, Lebail G, Chollet-Xemard C, Maxime V, Brun-Buisson C, Lefrant JY, Bollaert PE, Megarbane B, Ricard JD, Anguel N, Vicaut E, Adnet F; KETASED Collaborative Study Group. Etomidate versus ketamine for rapid sequence intubation in acutely ill patients: a multicentre randomised controlled trial. Lancet. 2009 Jul 25;374(9686):293-300. doi: 10.1016/S0140-6736(09)60949-1. Epub 2009 Jul 1. PMID 19573904
- [Background] Hinkewich C, Green R. The impact of etomidate on mortality in trauma patients. Can J Anaesth. 2014 Jul;61(7):650-5. doi: 10.1007/s12630-014-0161-6. Epub 2014 Apr 11. PMID 24723214
- [Background] Hohl CM, Kelly-Smith CH, Yeung TC, Sweet DD, Doyle-Waters MM, Schulzer M. The effect of a bolus dose of etomidate on cortisol levels, mortality, and health services utilization: a systematic review. Ann Emerg Med. 2010 Aug;56(2):105-13.e5. doi: 10.1016/j.annemergmed.2010.01.030. Epub 2010 Mar 25. PMID 20346542
- [Background] McPhee LC, Badawi O, Fraser GL, Lerwick PA, Riker RR, Zuckerman IH, Franey C, Seder DB. Single-dose etomidate is not associated with increased mortality in ICU patients with sepsis: analysis of a large electronic ICU database. Crit Care Med. 2013 Mar;41(3):774-83. doi: 10.1097/CCM.0b013e318274190d. PMID 23318491
- [Background] Warner KJ, Cuschieri J, Jurkovich GJ, Bulger EM. Single-dose etomidate for rapid sequence intubation may impact outcome after severe injury. J Trauma. 2009 Jul;67(1):45-50. doi: 10.1097/TA.0b013e3181a92a70. PMID 19590307
- [Background] Upchurch CP, Grijalva CG, Russ S, Collins SP, Semler MW, Rice TW, Liu D, Ehrenfeld JM, High K, Barrett TW, McNaughton CD, Self WH. Comparison of Etomidate and Ketamine for Induction During Rapid Sequence Intubation of Adult Trauma Patients. Ann Emerg Med. 2017 Jan;69(1):24-33.e2. doi: 10.1016/j.annemergmed.2016.08.009. PMID 27993308
- [Background] Fields AM, Rosbolt MB, Cohn SM. Induction agents for intubation of the trauma patient. J Trauma. 2009 Oct;67(4):867-9. doi: 10.1097/TA.0b013e3181b021c5. No abstract available. PMID 19820598
- [Background] Baird CR, Hay AW, McKeown DW, Ray DC. Rapid sequence induction in the emergency department: induction drug and outcome of patients admitted to the intensive care unit. Emerg Med J. 2009 Aug;26(8):576-9. doi: 10.1136/emj.2008.067801. PMID 19625554
- [Background] Zettervall SL, Sirajuddin S, Akst S, Valdez C, Golshani C, Amdur RL, Sarani B, Dunne JR. Use of propofol as an induction agent in the acutely injured patient. Eur J Trauma Emerg Surg. 2015 Aug;41(4):405-11. doi: 10.1007/s00068-014-0479-3. Epub 2014 Nov 20. PMID 26038005
- [Background] Choi YF, Wong TW, Lau CC. Midazolam is more likely to cause hypotension than etomidate in emergency department rapid sequence intubation. Emerg Med J. 2004 Nov;21(6):700-2. doi: 10.1136/emj.2002.004143. PMID 15496697
- [Background] Morris C, Perris A, Klein J, Mahoney P. Anaesthesia in haemodynamically compromised emergency patients: does ketamine represent the best choice of induction agent? Anaesthesia. 2009 May;64(5):532-9. doi: 10.1111/j.1365-2044.2008.05835.x. PMID 19413824
- [Background] Miller M, Kruit N, Heldreich C, Ware S, Habig K, Reid C, Burns B. Hemodynamic Response After Rapid Sequence Induction With Ketamine in Out-of-Hospital Patients at Risk of Shock as Defined by the Shock Index. Ann Emerg Med. 2016 Aug;68(2):181-188.e2. doi: 10.1016/j.annemergmed.2016.03.041. Epub 2016 Apr 27. PMID 27130803
- [Background] Lyon RM, Perkins ZB, Chatterjee D, Lockey DJ, Russell MQ; Kent, Surrey & Sussex Air Ambulance Trust. Significant modification of traditional rapid sequence induction improves safety and effectiveness of pre-hospital trauma anaesthesia. Crit Care. 2015 Apr 1;19(1):134. doi: 10.1186/s13054-015-0872-2. PMID 25879683
- [Background] Kolenda H, Gremmelt A, Rading S, Braun U, Markakis E. Ketamine for analgosedative therapy in intensive care treatment of head-injured patients. Acta Neurochir (Wien). 1996;138(10):1193-9. doi: 10.1007/BF01809750. PMID 8955439
- [Background] Bourgoin A, Albanese J, Wereszczynski N, Charbit M, Vialet R, Martin C. Safety of sedation with ketamine in severe head injury patients: comparison with sufentanil. Crit Care Med. 2003 Mar;31(3):711-7. doi: 10.1097/01.CCM.0000044505.24727.16. PMID 12626974
- [Background] Hughes S. Towards evidence based emergency medicine: best BETs from the Manchester Royal Infirmary. BET 3: is ketamine a viable induction agent for the trauma patient with potential brain injury. Emerg Med J. 2011 Dec;28(12):1076-7. doi: 10.1136/emermed-2011-200891. PMID 22101599
- [Result] Bergen JM, Smith DC. A review of etomidate for rapid sequence intubation in the emergency department. J Emerg Med. 1997 Mar-Apr;15(2):221-30. doi: 10.1016/s0736-4679(96)00350-2. PMID 9144065
- [Result] Pillay L, Hardcastle T. Collective Review of the Status of Rapid Sequence Intubation Drugs of Choice in Trauma in Low- and Middle-Income Settings (Prehospital, Emergency Department and Operating Room Setting). World J Surg. 2017 May;41(5):1184-1192. doi: 10.1007/s00268-016-3712-x. PMID 27646281
- [Result] Mayglothling J, Duane TM, Gibbs M, McCunn M, Legome E, Eastman AL, Whelan J, Shah KH; Eastern Association for the Surgery of Trauma. Emergency tracheal intubation immediately following traumatic injury: an Eastern Association for the Surgery of Trauma practice management guideline. J Trauma Acute Care Surg. 2012 Nov;73(5 Suppl 4):S333-40. doi: 10.1097/TA.0b013e31827018a5. PMID 23114490
- [Result] Ballow SL, Kaups KL, Anderson S, Chang M. A standardized rapid sequence intubation protocol facilitates airway management in critically injured patients. J Trauma Acute Care Surg. 2012 Dec;73(6):1401-5. doi: 10.1097/TA.0b013e318270dcf5. PMID 23188232